CLINICAL TRIAL: NCT01295294
Title: International, Prospective, Double-blind, 3-arm Comparative, Randomized, Placebo-controlled Phase IV Study on the Effect of Counseling and Either Tranexamic Acid or Mefenamic Acid or Placebo, on the Management of Bleeding/Spotting in Women Using the Levonorgestrel-releasing Intrauterine System (MIRENA) for Contraception.
Brief Title: Management of Initial Bleeding/Spotting Associated With the Levonorgestrel-releasing Intrauterine System (MIRENA)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15105; 2010-020922-16 (EudraCT Number)
Record Dates: First submitted 2011-02-11; First posted 2011-02-14 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-11

CONDITIONS: Uterine Hemorrhage
Keywords: Uterine Hemorrhage; Contraception; Contraceptive Methods; Intrauterine devices; Mirena
MeSH Terms: conditions — Uterine Hemorrhage | interventions — Tranexamic Acid; Mefenamic Acid; Levonorgestrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- tranexamic acid + Mirena (Levonorgestrel IUS, BAY86-5028) (Experimental): Subjects with successful MIRENA insertion will receive treatments with tranexamic acid
  Interventions: Drug: Tranexamic acid; Drug: Mirena (Levonorgestrel IUS, BAY86-5028)
- mefenamic acid + Mirena (Levonorgestrel IUS, BAY86-5028) (Experimental): Subjects with successful MIRENA insertion will receive treatments with mefenamic acid
  Interventions: Drug: Mefenamic acid; Drug: Mirena (Levonorgestrel IUS, BAY86-5028)
- placebo + Mirena (Levonorgestrel IUS, BAY86-5028) (Placebo Comparator): Subjects with successful MIRENA insertion will receive placebo
  Interventions: Drug: Placebo; Drug: Mirena (Levonorgestrel IUS, BAY86-5028)

INTERVENTIONS:
Drug: Tranexamic acid — 500 mg 3 times daily per oral during bleeding/spotting episodes
  Arms: tranexamic acid + Mirena (Levonorgestrel IUS, BAY86-5028)
Drug: Mefenamic acid — 500 mg 3 times daily per oral during bleeding/spotting episodes
  Arms: mefenamic acid + Mirena (Levonorgestrel IUS, BAY86-5028)
Drug: Placebo — 3 times daily per oral during bleeding/spotting episodes
  Arms: placebo + Mirena (Levonorgestrel IUS, BAY86-5028)
Drug: Mirena (Levonorgestrel IUS, BAY86-5028) — In vitro release rate 20 microgram/24 hours. Intrauterine system

SUMMARY:
The purpose of the study is to investigate if the study drugs (tranexamic acid or mefenamic acid) can control irregular bleeding during the first 3 months of using Mirena. The study drugs tested are tested against placebo ("dummy medication not containing any active drug"). Treatment period is followed by a one-month period when study drugs are not taken but Mirena use is continued.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent
* Healthy female subjects requesting contraception
* Age: 18 - 45 years inclusive
* Successful interval insertion of MIRENA
* History of regular cyclic menstrual periods
* Normal or clinically insignificant cervical smear not requiring further follow up

Exclusion Criteria:

* Pregnancy or lactation
* Climacteric symptoms prior to the screening visit
* Known or suspected clinically significant ovarian cysts, endometrial polyps, fibroids, or other genital organ pathology, that, in the opinion of the investigator, may interfere with the assessment of the bleeding profile during the study
* Undiagnosed abnormal genital bleeding
* Current or history of thrombembolic disease, or established risk factors for venous thromboembolism
* Current migraine, focal migraine with asymmetrical visual loss or other symptoms indicating transient cerebral ischemia, or exceptionally severe headaches
* Hypersensitivity to any ingredient of the investigational medicinal products or the non-investigational medicinal product
* Daily or frequent use of a nonsteroidal anti-inflammatory drug (NSAIDs) for any condition
* Not willing to use nonsteroidal anti-inflammatory drug (NSAIDs) medication as pain medication during the double blind treatment period

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 187 (Actual)
Dates: Start 2011-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
The primary efficacy variable will be the cumulative number of bleeding / spotting days | During 90 day double-blind treatment period

SECONDARY OUTCOMES:
To describe and compare the bleeding patterns observed in women during treatment period | 90 day treatment period
To describe and compare the bleeding patterns observed in women during follow-up period | During the 30 day follow-up period
Satisfaction with oral blinded study drug treatment for bleeding / spotting | 90 day treatment period
Occurrence of dysmenorrhea | During 120 day study period
Continuation rate with study drug | During the 90 day treatment period
Continuation rate with Mirena | During 120 day study period
Adverse Events Collection | Until day 120
Number of spotting-only days | During the 90-day treatment period
Number of bleeding / spotting episodes | During the 90-day treatment period
Length of bleeding / spotting episodes | During the 90-day treatment period
Number of bleeding days with heavy intensity | During the 90-day treatment period
Change in the number of B/S days between Day 60 and Day 90 of MIRENA use and the 30-day follow-up period | Up to day 120
Satisfaction with levonorgestrel-releasing intrauterine system | Up to day 120
Number of days of pain medication for dysmenorrhea during the 90 day treatment period | During the 90-day treatment period
Number of bleeding-only days | During the 90-day treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (12):
- Denmark (6):
  - Aalborg
  - Århus C
  - København NV
  - Odense C
  - Skive
  - Søborg
- Ireland (3):
  - Mallow, Cork
  - Blackrock, Dublin
  - Cork
- Norway (3):
  - Elverum
  - Haugesund
  - Trondheim

REFERENCES:
- [Derived] Sordal T, Inki P, Draeby J, O'Flynn M, Schmelter T. Management of initial bleeding or spotting after levonorgestrel-releasing intrauterine system placement: a randomized controlled trial. Obstet Gynecol. 2013 May;121(5):934-941. doi: 10.1097/AOG.0b013e31828c65d8. PMID 23635728
- See also: Click here and search for information of Bayer products for Europe — http://www.clinicaltrialsregister.eu